CLINICAL TRIAL: NCT01917890
Title: Radiation Therapy With or Without Curcumin Supplement in Treating Patients With Prostate Cancer
Brief Title: Radiosensitizing and Radioprotectve Effects of Curcumin in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Rastmanesh, Dr., Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Radiation Therapy And Curcumin
Record Dates: First submitted 2013-08-03; First posted 2013-08-07 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer; Radiation Therapy
Keywords: curcumin; radioprotective; radiosensitizer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin Group (Experimental): Patients undergo 74 Gy of intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Patients take 3 grams of curcumin (as 6 capsules 500 mg)
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): Patients undergo 74 Gy of intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Patients take 3 grams of placebo (as 6 capsules 500 mg)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Patients undergo 74 Gy of intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Patients take 3 grams of BCM95 Curcumin (as 6 × 500 mg capsules)
  Other Names: turmeric pigment
  Arms: Curcumin Group
Dietary Supplement: Placebo — Patients undergo 74 Gy of intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Patients take 3 grams of roasted rice powder (as 6 × 500 mg capsules)
  Arms: Placebo

SUMMARY:
Prostate cancer is the second most incident cancer among male population worldwide. Radiation therapy by itself or along with surgery and chemotherapy are the main treatments for prostate cancer however prostate cancer cells are only modestly responsive or even unresponsive to the cytotoxic effects of radiotherapy. Recently some in vitro and in vivo studies showed radiosensitizing and radioprotective effects for curcumin. No clinical trial has been done in this area and it is not yet known whether radiation therapy is more effective with or without curcumin supplements in treating patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. Age range of 50-80
3. ECOG performance status 0-1
4. Life expectancy > 5 years
5. Must be enrolled in a social security program
6. No other cancer, except basal cell skin cancer, that has been treated or relapsed within the past 5 years
7. No severe uncontrolled hypertension (systolic BP ≥ 160 mm Hg or diastolic BP ≥ 90 mm Hg)
8. No contraindication to luteinizing hormone-releasing hormone agonists
9. No contraindication to pelvic irradiation (e.g., scleroderma, chronic inflammatory gastrointestinal disease)
10. No hip prosthesis
11. Must not be deprived of liberty or under guardianship
12. No geographical, social, or psychological reasons that would preclude follow up

Exclusion Criteria:

1. Clinical stage T3 or T4
2. Gleason score ≥ 8
3. Serum PSA ≥ 20 ng/mL and ≤ 100 ng/mL
4. other prior surgery for prostate cancer
5. concurrent participation in another clinical trial which would require approval upon entry to this trial
6. Gastrointestinal disorders such as IBD, reflux and peptic ulcers
7. Any adverse reaction to curcumin

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Biochemical or clinical progression-free survival | 1 year
  To assess this outcome the results of magnetic resonance spectroscopy (MRS)will be compared between the 2 groups 1 week before radiation therapy and 3 months after radiotherapy completion. Also prostate specific antigen (PSA)rebound will be compared between the 2 groups after 1 year. Side effects of treatment during 1 year after treatment completion will be compared between the 2 groups using questionnaires and physical examination

SECONDARY OUTCOMES:
Quality of life | 1 year
  Quality of life related issues will be compared between the 2 groups 1 week before radiotherapy onset and 3 months and 1 year after radiotherapy completion using EORTC QLQ-C30 and EORTC QLQ - PR25
Sexual dysfunction score | 1 year
  Sexual dysfunction score will be compared between the 2 groups 1 week before radiotherapy onset and 3 months and 1 year after radiotherapy completion using EORTC QLQ - PR25
C-reactive protein (hs-CRP) | 5 months
  It will be measured in plasma 1 week before radiotherapy onset and 3 month after radiotherapy completion using biochemical kits. (mg/L)
Inflammatory factors (tumor necrosis factor alpha (TNF-alpha), Interleukin 1 beta (IL1-beta)and Interleukin 6 (ILl-6)) | 5 monthes
  They will be measured in plasma 1 week before radiotherapy onset and 3 month after radiotherapy completion using biochemical kits. (pg/ml)
Antioxidant enzymes (Catalase, super oxide dismutase (SOD), glutathione-S- transferase (GST), glutathione peroxidase (GPX)) | 5 months
  They will be measured in plasma 1 week before radiotherapy onset and 3 month after radiotherapy completion using biochemical kits. (U/L)
cycloxygenase 2 (COX2) | 5 months
  measuring activity and gene expression of the enzyme in peripheral blood mono-nuclear cell (PBMC)1 week before radiotherapy onset and 3 months after radiotherapy.
Nuclear factor KB (NF-ΚB) | 5 months
  measuring activity and gene expression in peripheral blood mono-nuclear cell (PBMC)1 week before radiotherapy onset and 3 months after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rastmanesh, PhD, Study Chair — Clinical Nutrition & Dietetics Dept., Shahid Beheshti University of Medical Sciences,
Locations (1):
- Oncology and radiotherapy department, Besat Hospital, Tehran, Tehran Province, Iran